CLINICAL TRIAL: NCT01232738
Title: A Multi-Center Controlled Screening Trial of Safety and Efficacy of Rasagiline in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Trial of Safety and Efficacy of Rasagiline in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yunxia Wang, MD (Other)
Collaborators: Western ALS Study Group (Unknown)
Responsible Party: Sponsor-Investigator, Yunxia Wang, MD, Assistant Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11922
Record Dates: First submitted 2010-10-22; First posted 2010-11-02 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — rasagiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rasagiline (Experimental): Treated for 12 months with rasagiline 2mg orally, once daily.
  Interventions: Drug: rasagiline

INTERVENTIONS:
Drug: rasagiline — rasagiline 2 mg daily for 12 months

SUMMARY:
ALS is a disorder that weakens motor strength and lung function. Rapid loss of motor neurons in the brain and spinal cord of ALS patients causes the symptoms of increasing weakness and loss of muscle function. While there are drugs to help relieve symptoms of ALS, there is no cure for ALS.

Rasagiline is a drug with possible neuroprotective characteristics. Neuroprotective means that the nervous system may be protected against weakening. It is known that rasagiline has possible neuroprotective characteristics and it is approved for use for patients with another disorder, the effectiveness of rasagiline for patients with ALS has not been tested.

DETAILED DESCRIPTION:
The specific aim of this screen study is to determine whether rasagiline is safe in this patient population and if the drug has the potential to slow ALS disease progression

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of laboratory-supported probable, probable, or definite ALS, according to a modified El Escorial criteria, by the study investigator (Appendix IV).
2. 21 to 80 years of age inclusive.
3. VC greater or equal to 75% of predicted at screening and baseline.
4. Onset of weakness within 3 years prior to enrollment.
5. If patients are taking riluzole for ALS, they must be on a stable dose for at least thirty days prior to the baseline visit.
6. Women of childbearing age must be non-lactating and surgically sterile or using an effective method of birth control and have a negative pregnancy test.
7. Willing and able to give signed informed consent that has been approved by the Institutional Review Board (IRB).

Exclusion criteria

1. Requirement for tracheotomy ventilation or non-invasive ventilation for > 23 hours per day.
2. Patients on sympathomimetic agents. This includes pseudoephedrine, phenylephrine, phenylpropanolamine, and ephedrine.
3. Patients on analgesics with serotoninergic properties such as meperidine, tramadol, methadone and propoxyphen, flexeril.
4. Patients on fluoxetine or fluvoxamine.
5. Patients taking amitriptyline > 50 mg/d, trazodone and sertraline > 100 mg/d, citalogram > 20 mg/d or paroxetine > 30 mg/d.
6. Diagnosis of other neurodegenerative diseases (Parkinson disease, Alzheimer disease, etc).
7. Clinically significant history of unstable medical illness (unstable angina, advanced cancer, etc) over the last 30 days.
8. History of renal disease.
9. History of liver disease.
10. Current pregnancy or lactation.
11. Limited mental capacity such that the patient cannot provide written informed consent or comply with evaluation procedures.
12. History of recent alcohol or drug abuse or noncompliance with treatment or other experimental protocols.
13. VC < 75% of predicted.
14. Receipt of any investigational drug within the past 30 days.
15. Women with the potential to become pregnant who are not practicing effective birth control.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yunxia Wang, MD, Principal Investigator — University of Kansas Medical Center
Locations (10):
- United States (9):
  - Phoenix Neurological Institute, Phoenix, Arizona
  - California Pacific Medical Center, San Francisco, California
  - University of Iowa, Iowa City, Iowa
  - University Of Kansas Medical Center, Kansas City, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
  - The Methodist Hospital System, Houston, Texas
- McGill University, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Rasagiline: Open label study of rasagiline at 2 mg daily for 12 months
Period: Overall Study
Arm/Group | Rasagiline
Started | 36
Completed | 23
Not Completed | 13
Not completed — Death | 3
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Groups:
- Rasagiline: Open label study of 2 mg rasagiline daily
Arm/Group | Rasagiline
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 17
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R)
Description: The primary outcome measure is the difference in the rate of decline in function, as detected by the ALS Functional Rating Scale - Revised (ALSFRS-R) in patients taking rasagiline compared to a database of patients from randomized clinical trials conducted during 1997-2007. Minimum score is 0 (no function) to Maximum score is 48 (normal function)
Time Frame: up to 12 months
Population: The placebo arm are from the randomized, controlled studies in ALS performed during 2004-2010, corrected for symptom duration.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- ALSRFS-R Slope - Rasagiline: Change in ALSRFS-R at 12 months
- ALSFRS-R - Historical Placebo Control: Change in slope in the Historical Placebo Control group
Arm/Group | ALSRFS-R Slope - Rasagiline | ALSFRS-R - Historical Placebo Control
Number analyzed (Participants) | 36 | 478
units on a scale | -1.20 (0.14) | -0.94 (0.04)
Statistical Analysis 1: Comparison: ALSRFS-R Slope - Rasagiline vs ALSFRS-R - Historical Placebo Control; Difference in slope of decline; Test type: Superiority; p = 0.07, Chi-squared; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.53 to 0.02]

2. Secondary Outcome: Difference in Time to Treatment Failure
Description: This group is defined as death, endotracheal intubation, tracheostomy-assisted ventilation or use of noninvasive ventilation >= 23 hours/day for 14 days or more.
Time Frame: up to 12 months
Population: Failure was defined as death, endotracheal intubation, tracheostomy-assisted ventilation, or use of noninvasive ventilation 23 hours/day for 14 days or more. It is defined in years.
Measure: Median (95% Confidence Interval); unit: years
Groups:
- Difference in Time to Treatment Failure - Rasagiline: This group is defined as death, endotracheal intubation, tracheostomy-assisted ventilation or noninvasive ventilation >=23 hours/day for 14 days.
- Difference in Time to Treatment Failure - Historical Control: Historical Controls were from the previous ALS trials.
Arm/Group | Difference in Time to Treatment Failure - Rasagiline | Difference in Time to Treatment Failure - Historical Control
Number analyzed (Participants) | 36 | 203
years | 0.9367 [0.7682 to 0.9839] | 0.8963 [0.8438 to 0.9318]
Statistical Analysis 1: Comparison: Difference in Time to Treatment Failure - Rasagiline vs Difference in Time to Treatment Failure - Historical Control; Test type: Superiority; p = 0.58, Log Rank

3. Other Pre Specified Outcome: Change in JC-1 Mitochondrial Biomarkers
Description: The 12 month change in mitochondrial biomarkerJC-1 red/green fluorescence ratio. We measured at baseline, 6 months and 12 months.
Time Frame: Baseline, 6 months, 12 months
Population: Only 14 subjects that completed the study were able to have this biomarker analyzed.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Rasagiline
Number analyzed (Participants) | 14
ratio | 1.92 [1.14 to 2.70]

4. Other Pre Specified Outcome: Change in Mitotracker Mitochondrial Biomarkers
Description: The 12 month change in mitochondrial biomarkerMitotracker. We measured at baseline, 6 months and 12 months.
Time Frame: Baseline, 6 months, 12 months
Population: Only 17 subjects that completed the study were able to have this biomarker analyzed.
Measure: Mean (95% Confidence Interval); unit: Relative Fluorescent Intensity
Arm/Group | Rasagiline
Number analyzed (Participants) | 17
Relative Fluorescent Intensity | 54.14 [31.47 to 76.81]

5. Other Pre Specified Outcome: Change in Percent Annexin V Mitochondrial Biomarkers
Description: The 12 month change in mitochondrial biomarker Annexin V %. We measured at baseline, 6 months and 12 months.
Time Frame: Baseline, 6 months, 12 months
Population: Only 17 subjects that completed the study were able to have this biomarker analyzed.
Measure: Mean (95% Confidence Interval); unit: Annexin V %
Arm/Group | Rasagiline
Number analyzed (Participants) | 17
Annexin V % | -6.67 [-20.3 to 6.7]

6. Other Pre Specified Outcome: Change in BCL2/BAX Mitochondrial Biomarkers
Description: The 12 month change in mitochondrial biomarker BCL2/BAX. We measured at baseline, 6 months and 12 months.
Time Frame: Baseline, 6 months, 12 months
Population: Only 10 subjects that completed the study were able to have this biomarker analyzed.
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Rasagiline
Number analyzed (Participants) | 10
Ratio | 0.24 [0.24 to 0.27]

7. Other Pre Specified Outcome: Change in ORAC Mitochondrial Biomarkers
Description: The 12 month change in mitochondrial biomarker Oxygen Radical Antioxidant Capacity. We measured at baseline, 6 months and 12 months.
Time Frame: Baseline, 6 months, 12 months
Population: Only 17 subjects that completed the study were able to have this biomarker analyzed.
Measure: Mean (95% Confidence Interval); unit: Trolox equivalents
Arm/Group | Rasagiline
Number analyzed (Participants) | 17
Trolox equivalents | 1028.70 [681.09 to 1376.31]

8. Other Pre Specified Outcome: Change in ORAC Mitochondrial Biomarkers
Description: as for outcome 7
Time Frame: Baseline, 6 months, 12 months
Population: Only 17 subjects that completed the study were able to have this biomarker analyzed.
Measure: Mean (95% Confidence Interval); unit: umol Trolox equivalents
Arm/Group | Rasagiline
Number analyzed (Participants) | 17
umol Trolox equivalents | 1028.70 [681.09 to 1376.31]

9. Other Pre Specified Outcome: Change in ORAC Mitochondrial Biomarkers
Description: as for outcome 7
Time Frame: Baseline, 6 months, 12 months
Population: Only 17 subjects that completed the study were able to have this biomarker analyzed.
Measure: Mean (95% Confidence Interval); unit: Trolox equivalents
Arm/Group | Rasagiline
Number analyzed (Participants) | 17
Trolox equivalents | 1028.70 [681.09 to 1376.31]

ADVERSE EVENTS:
Arm/Group | Rasagiline
Serious Adverse Events (participants affected / at risk) | 1/36
Other Adverse Events (participants affected / at risk) | 17/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rasagiline (N=36)
Fracture (Injury, poisoning and procedural complications) | 1 (1) — Fractured pelvic bone
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rasagiline (N=36)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Dizziness (Blood and lymphatic system disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Hypertension (Blood and lymphatic system disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 4 (4)
Xerostomia (General disorders) | 1 (1)
Lab abnormality (elevated ALT) (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No